CLINICAL TRIAL: NCT05945901
Title: A Phase II/III, Double-blind, Randomized, Multi-center Study of HR070803 in Combination With Oxaliplatin, 5-fluorouracil, Calcium Folinate and Bevacizumab Versus FOLFOX in Combination With Bevacizumab for First-line Treatment of Advanced Colorectal Cancer
Brief Title: A Phase II/III Study of HR070803 in Combination With Oxaliplatin, 5-fluorouracil, Calcium Folinate and Bevacizumab Versus FOLFOX in Combination With Bevacizumab for First-line Treatment of Advanced Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR070803-306-CRC
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR070803 (Experimental): HR070803 plus oxaliplatin, 5-FU/LV, bevacizumab
  Interventions: Drug: HR070803 plus oxaliplatin, 5-FU/LV, bevacizumab
- HR070803 simulator (Placebo Comparator): HR070803 simulator plus oxaliplatin, 5-FU/LV, bevacizumab
  Interventions: Drug: HR070803 simulator plus oxaliplatin, 5-FU/LV, bevacizumab

INTERVENTIONS:
Drug: HR070803 plus oxaliplatin, 5-FU/LV, bevacizumab — HR070803 plus oxaliplatin, 5-FU/LV, bevacizumab Patients will receive the study drug after randomization, and those with effective efficacy evaluation (CR, PR or SD) will receive intravenous chemotherapy for up to 8-12 cycles, and then enter the maintenance treatment stage until PD, death, intolerable toxicity or withdrawal of informed consent (whichever occurs first)
  Arms: HR070803
Drug: HR070803 simulator plus oxaliplatin, 5-FU/LV, bevacizumab — HR070803 simulator plus oxaliplatin, 5-FU/LV, bevacizumab Patients will receive the study drug after randomization, and those with effective efficacy evaluation (CR, PR or SD) will receive intravenous chemotherapy for up to 8-12 cycles, and then enter the maintenance treatment stage until PD, death, intolerable toxicity or withdrawal of informed consent (whichever occurs first)
  Arms: HR070803 simulator

SUMMARY:
This is a double-blind, randomized, multi-center, II/III study in at least 606 patients with advanced colorectal cancer. The study is being conducted to evaluate the safety of HR070803 combined with oxaliplatin, 5-FU/LV and bevacizumab in phase II and to evaluate the efficacy of HR070803 in combination with oxaliplatin, 5-FU/LV, and bevacizumab versus HR070803 simulator in combination with FOLFOX and bevacizumab for first-line treatment of patients with unresectable metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female who is 18-75 years of age;
2. Histologically-confirmed metastatic and unresectable (Stage IV as defined by American Joint Committee on Cancer [AJCC eighth edition]) colorectal adenocarcinoma
3. No previous systemic antitumor therapy (including but not limited to systemic chemotherapy, molecularly targeted therapy, immunotherapy, biotherapy, and other investigational therapeutic agents) for colorectal cancer (patients with confirmed relapse ≥6 months after the last administration of neoadjuvant or adjuvant therapy can be enrolled);
4. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 ;
5. Life expectancy of ≥ 6 months;
6. Vital organ functions meet the criteria.

Exclusion Criteria:

1. With confirmed MMR deficient (dMMR) or microsatellite instability high (MSI-H).
2. With central nervous system metastases.
3. Previous oxaliplatin-containing chemotherapy within 12 months prior to enrolment.
4. Previous treatment with irinotecan, immune checkpoint inhibitor, anti-epidermal growth factor receptor or any anti-angiogenic drug.
5. Patients with large amount of pleural effusion, ascites or pericardial effusion that could not reach a stable state within 2 weeks prior to enrolment.
6. Severe gastrointestinal dysfunction (inflammation or diarrhea > grade 1).
7. With diagnosed interstitial lung disease.
8. Severe cardiovascular and cerebrovascular diseases.
9. Peripheral neuropathy > grade 1.
10. Intestinal obstruction within the 6 months prior to enrolment.
11. Gastrointestinal perforation, gastrointestinal fistula, intraperitoneal abscess, and non-gastrointestinal fistula (e.g. tracheoesophageal fistula) within 6 months prior to enrolment.
12. Patients with CTCAE≥ grade 3 gastrointestinal bleeding within 6 months prior to enrolment, or any grade gastrointestinal bleeding within 1 month prior to enrolment.
13. Patients with CTCAE≥ grade 3 extra-gastrointestinal bleeding within 6 months prior to enrolment, or CTCAE≥ grade 2 extra-gastrointestinal bleeding within 3 months prior to enrolment.
14. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg under regular antihypertensive therapy), and a history of hypertensive crisis or hypertensive encephalopathy.
15. History of hypersensitivity or contraindications to any of irinotecan liposomes/simulator, irinotecan, other liposomal products, 5-FU, calcium folinate, oxaliplatin, bevacizumab.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) According to NCI-CTCAE v5.0（Phase II） | From Baseline to primary completion date, about 48 months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant after signing the informed consent form and which does not necessarily have to have a causal relationship with this treatment. An AE could be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change infrequency and/or intensity) of a preexisting condition that is temporally associated with the use of study treatment, is also an AE.
Serious Adverse Events (SAE)（Phase II） | From Baseline to primary completion date, about 48 months
  An SAE is defined as any of the following adverse events in a participant or clinical investigation participant after signing the informed consent form and which does not necessarily have to have a causal relationship with this treatment: events that result in death, life-threatening events; events requiring hospitalization or prolonged hospitalization; events leading to permanent or severe disability/loss of function (significant impairment of the ability to carry out normal life functions); congenital abnormalities or birth defects; a medically important event or intervention may be required to prevent any of these outcomes.
Progression-Free Survival (PFS) Assessed by IRC（Phase III） | From Baseline to primary completion date, about 48 months
  from randomization to PD or death from any cause

SECONDARY OUTCOMES:
Overall Response Rate (ORR) Assessed by investigator（Phase II） | From Baseline to primary completion date, about 48 months
  The proportion of patients who acquired complete response and partial response during treatment.
Disease Control Rate (DCR) by investigator（Phase II） | From Baseline to primary completion date, about 48 months
  The proportion of patients who acquired complete response and partial response and stable disease during treatment.
Duration of Overall Response (DoR) by investigator（Phase II） | From Baseline to primary completion date, about 48 months
  For subjects who demonstrated CR or PR, response duration is defined as the time from the date of first response (CR or PR) until the date of first documented disease progression or death.
Progression-Free Survival (PFS) Assessed by investigator（Phase II） | From Baseline to primary completion date, about 48 months
  from randomization to PD or death from any cause.
Overall Survival (OS)（Phase II） | From Baseline to primary completion date, about 48 months
  from randomization to death from any cause.
Characterize the PK（Phase II） | From Baseline to primary completion date, about 48 months
  Serum concentrations of SN-38 and CPT-11 will be monitored. PK modeling will be performed and an appropriate model will be selected to describe the data.
Overall Survival (OS)（Phase III） | From Baseline to primary completion date, about 48 months
  from randomization to death from any cause.
Progression-Free Survival (PFS) Assessed by investigator（Phase III） | From Baseline to primary completion date, about 48 months
  from randomization to PD or death from any cause.
Overall Response Rate (ORR) Assessed by IRC and investigator（Phase III） | From Baseline to primary completion date, about 48 months
  The proportion of patients who acquired complete response and partial response during treatment.
Duration of Overall Response (DoR) by IRC and investigator（Phase III） | From Baseline to primary completion date, about 48 months
  For subjects who demonstrated CR or PR, response duration is defined as the time from the date of first response (CR or PR) until the date of first documented disease progression or death.
Disease Control Rate（DCR） by IRC and investigator（Phase III） | From Baseline to primary completion date, about 48 months
  The proportion of patients who acquired complete response and partial response and stable disease during treatment.
Adverse Events (AE) According to NCI-CTCAE v5.0（Phase III） | From Baseline to primary completion date, about 48 months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant after signing the informed consent form and which does not necessarily have to have a causal relationship with this treatment. An AE could be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change infrequency and/or intensity) of a preexisting condition that is temporally associated with the use of study treatment, is also an AE.
Serious Adverse Events (SAE)（Phase III） | From Baseline to primary completion date, about 48 months
  An SAE is defined as any of the following adverse events in a participant or clinical investigation participant after signing the informed consent form and which does not necessarily have to have a causal relationship with this treatment: events that result in death; life-threatening events; events requiring hospitalization or prolonged hospitalization; events leading to permanent or severe disability/loss of function (significant impairment of the ability to carry out normal life functions); congenital abnormalities or birth defects; a medically important event or intervention may be required to prevent any of these outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdog, China

IPD SHARING:
Plan to Share IPD: Undecided